CLINICAL TRIAL: NCT00466973
Title: Randomized Comparison of Ablation Devices Used During Surgery for the Treatment of Atrial Fibrillation
Brief Title: Atrial Fibrillation Ablation Device Comparison Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/11/VA07
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; ablation device comparison; ablation in right atria
MeSH Terms: conditions — Atrial Fibrillation | interventions — Constriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dry bipolar radiofrequency (RF) clamp (Active Comparator): used for ablation during surgical procedure
  Interventions: Device: Dry bipolar radiofrequency (RF) clamp
- Unipolar microwave antenna (Active Comparator): used for ablation during surgical procedure
  Interventions: Device: Unipolar microwave antenna
- Unipolar cryothermic probe (Active Comparator): used for ablation during surgical procedure
  Interventions: Device: Unipolar cryothermic probe
- Irrigated unipolar RF antenna (Active Comparator): used for ablation during surgical procedure
  Interventions: Device: Irrigated unipolar RF antenna
- Irrigated bipolar RF clamp (Active Comparator): used for ablation during surgical procedure
  Interventions: Device: Irrigated bipolar RF clamp
- Hi-intensity focused ultrasound wand (Active Comparator): used for ablation during surgical procedure
  Interventions: Device: Hi-intensity focused ultrasound wand

INTERVENTIONS:
Device: Dry bipolar radiofrequency (RF) clamp — Specified device used for ablation during standard surgical procedure
  Other Names: AtriCure
  Arms: Dry bipolar radiofrequency (RF) clamp
Device: Unipolar microwave antenna — Specified device used for ablation during standard surgical procedure
  Other Names: Boston Scientific FLEX 10
  Arms: Unipolar microwave antenna
Device: Unipolar cryothermic probe — Specified device used for ablation during standard surgical procedure
  Other Names: Cryocath SurgiFrost
  Arms: Unipolar cryothermic probe
Device: Irrigated unipolar RF antenna — Specified device used for ablation during standard surgical procedure
  Other Names: ESTECH Cobra Adhere
  Arms: Irrigated unipolar RF antenna
Device: Irrigated bipolar RF clamp — Specified device used for ablation during standard surgical procedure
  Other Names: Meditronic Cardioblate BP
  Arms: Irrigated bipolar RF clamp
Device: Hi-intensity focused ultrasound wand — Specified device used for ablation during standard surgical procedure
  Other Names: St. Jude Epicor
  Arms: Hi-intensity focused ultrasound wand

SUMMARY:
Atrial fibrillation is an irregular heart rhythm which requires long term anticoagulation to prevent risk of stroke and long term poor outcomes. At the same time one have heart surgery, a small additional procedure can be done to treat atrial fibrillation. Surgeons have a choice of six different devices that he or she can use to treat your atrial fibrillation. It is not known at this point which device is best at treating you, as each device seems to have the same success rate at curing atrial fibrillation. One of the six devices will be selected randomly by card pulled out at the time of enrollment. It is therefore the purpose of this study to compare the devices to each other and to follow up after surgery to determine if any one device is best. This information will be valuable to surgeons and to patients as the treatment for atrial fibrillation develops in the future.

DETAILED DESCRIPTION:
Surgery has been used as a treatment for atrial fibrillation (AF) for more than 20 years. Although highly successful, it has not been widely adopted because operations designed to cure AF require extensive cutting and suturing of the heart, inflicting a significant risk on the patient. Newer technologies now permit the surgeon to create similar scars on the heart as cutting, but much more quickly and safely than before.

Over the last ten years at least six different devices have been developed, each of which can scar the heart: Microwave, radiofrequency, ultrasound, laser and cold are some of them. Although there are many papers in the literature studying these devices, each seems to cure about 80% of patients with very low risk of morbidity and/or mortality. This leaves the surgeon with almost no basis upon which to base his or her selection of a device: Which is the best? Which should be used? Therefore, a comparison study is like this is desperately needed.

At the time of the surgery, surgeon who perform the AF treatment, he or she will select one of the six devices mentioned above at randomly assigned earlier, at the time of the enrollment. The device will be used to make scars on your heart exactly as described in the manufacturer's instructions and according to the surgeon's experience. The operation will then be completed per routine. In other words, the only part of the procedure that will be done differently from any other is that the actual device chosen to perform the ablation will vary from one study subject to another.

Patients will be followed up upto one year with EKGs, Holter monitors, MRI's, 6 minute walk tests, echocardiograms, blood tests like bNP and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing concomitant cardiac surgery who also have AF.

Exclusion Criteria:

* Patients undergoing re-do or emergency procedures
* Females of child-bearing age who are pregnant
* Age less than 19 and more than 75 years old

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11-20 (Actual); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial fibrillation | 3 months after surgery
  No atrial fibrillation noted by standard testing (Spot ECG, history, 24-hour Holter recording, Cardiac MRI or echocardiogram, Brain Natriuretic Peptide (BNP) levels
Rhythm at 12 months | 12 months after surgery
  No atrial fibrillation noted by standard testing (Spot ECG, history, 24-hour Holter recording, Cardiac MRI or echocardiogram, BNP levels
Major Adverse Cardiovascular Events (MACEs) at 1 and 3 months | 1 and 3 months post-surgical procedure
  Recording any major adverse cardiovascular events reported

SECONDARY OUTCOMES:
Functional and qualitative improvement in heart failure, ejection fraction, left atrial size, exercise tolerance | 6 and 12 months post-surgical procedure
  Quality of life questionnaire
Rhythm at 3, 6 and 9 months | 3, 6 and 9 months post-surgical procedure
  No atrial fibrillation noted by standard testing (Spot ECG, history, 24-hour Holter recording, Cardiac MRI or echocardiogram, BNP levels
All other adverse events | From surgical procedure through 12 months follow-up
  Any adverse events noted throughout period

CONTACTS AND LOCATIONS:
Overall Officials: Adam E Saltman, MD, Principal Investigator — Director Atrial fibrillation Program, Cardiothoracic Surgeon; Kamran B Ali, MD, Principal Investigator — Cardiology Fellow
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States